CLINICAL TRIAL: NCT01004965
Title: Multidrug Resistance Studies in Acute Myeloid Leukemia
Brief Title: Study of Bone Marrow and Blood Samples in Patients With Untreated Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia Enrolled on Clinical Trial CALGB-9621 or CALGB-9720
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9760; U10CA031946 (NIH); CALGB-9760; CDR0000078568 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Leukemia
Keywords: untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Samples are obtained: 1) pretreatment, 2) at the time of documentation of refractory disease in acute myeloid leukemia (AML) patients who do not achieve complete response (CR) after induction therapy, and 3) at the time of first relapse in patients who achieve CR.
  Marrow cells are preferentially used for all samples, but peripheral blood is acceptable if marrow is not available and the blood contains 20% or more blasts.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
This research study is looking at bone marrow and blood samples in patients with untreated acute myeloid leukemia or acute lymphoblastic leukemia enrolled on clinical trial CALGB-9621, CALGB-9720, CALGB 19808, and CALGB 10201. Studying samples of bone marrow and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine Pgp antigen expression and Pgp-mediated functional multidrug resistance (MDR) in pretreatment acute myeloid leukemia (AML) cells from adult patients enrolled on CALGB clinical trials of PSC-833 Pgp modulation.

II. Correlate Pgp-mediated MDR with patient pretreatment characteristics including age, immunophenotype, and karyotype.

III. Correlate Pgp expression, function, and in vitro modulation by PSC-833 with treatment outcome in previously untreated AML patients treated on CALGB Pgp modulation trials.

IV. Determine Pgp expression and function in AML cells from patients with refractory or relapsed leukemia following induction chemotherapy administered with or without PSC-833.

V. Correlate acquisition of drug resistance with changes in expression of other antigens and gain or loss of leukemic populations at relapse in these patients.

VI. Determine the role of other mediators, including multidrug resistance-associated protein (MRP) and lung-resistance protein (LRP), in mediating MDR in these patients at diagnosis and with relapsed or refractory disease after induction chemotherapy with or without PSC-833.

VII. Determine the frequency of Pgp-, MRP-, and LRP- mediated MDR in adult acute lymphoblastic leukemia cells and correlate this frequency with pretreatment characteristics and treatment outcome in these patients.

OUTLINE:

Samples are obtained: 1) pretreatment, 2) at the time of documentation of refractory disease in acute myeloid leukemia (AML) patients who do not achieve complete response (CR) after induction therapy, and 3) at the time of first relapse in patients who achieve CR.

Marrow cells are preferentially used for all samples, but peripheral blood is acceptable if marrow is not available and the blood contains 20% or more blasts. Pgp expression is measured using flow cytometry. AML samples are analyzed by immunoenzyme techniques (IET) using antibodies to CD33, CD34, and MRK16. B-lineage acute lymphoblastic leukemia (ALL) samples are analyzed by IET using antibodies to CD19, CD34, and MRK16. The antibodies used to analyze T-cells include CD7 and CD34. Pgp function is measured by growing cells in the presence of PSC-833 in vitro and then measuring Pgp expression as above. Multidrug resistance-associated protein (MRP) is measured using IET with the MRPm6 antibody. Lung-resistance protein (LRP) is measured with IET and the LRP56 antibody. These results are correlated with flow cytometry results.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients eligible for and registered to a CALGB multidrug resistance modulation treatment protocol for acute myeloid leukemia (CALGB 9621, CALGB-9720, CALGB-19808, and CALGB 10201) OR protocols for previously untreated acute lymphocytic leukemia
* Performance status: not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pateitns with acute myeloid leukemia enrolled on CALGB 9621, CALGB 9720, CALGB 19808 or CALGB 10201
Sampling Method: Non-Probability Sample
Enrollment: 2034 (Estimated)
Dates: Start 1997-03-15 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-06-16 (Actual)

PRIMARY OUTCOMES:
completion rate | Up to 5 years

SECONDARY OUTCOMES:
duration of completion rate | Up to 5 years
survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria R. Baer, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (46):
- United States (46):
  - Naval Medical Center - San Diego, San Diego, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - McLeod Regional Medical Center, Florence, South Carolina